CLINICAL TRIAL: NCT00065208
Title: Effects of Energy Healing on Prostate Cancer
Brief Title: Reiki/Energy Healing in Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Joan Fox, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001120 (NIH)
Record Dates: First submitted 2003-07-18; First posted 2003-07-22 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Reiki; Energy Healing
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutic Touch; Touch; RE1-silencing transcription factor; Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reiki (Experimental): Energy therapy
  Interventions: Behavioral: Reiki
- Pretend Reiki (Sham Comparator)
  Interventions: Behavioral: Pretend Reiki
- Rest / Guided Imagery (Other): Rest for pre-surgery outcomes Guided Imagery for post-surgery outcomes
  Interventions: Behavioral: Rest / Guided Imagery

INTERVENTIONS:
Behavioral: Reiki — Energy therapy - 8 biweekly sessions of 30 minutes
  Other Names: Energy Therapy; Touch Therapy; Energy Healing
  Arms: Reiki
Behavioral: Pretend Reiki — Touch from untrained pretend practitioners. 8 biweekly sessions of 30 minutes
  Other Names: Touch
  Arms: Pretend Reiki
Behavioral: Rest / Guided Imagery — 4 weekly sessions of 30 supine rest listening to soft music. One session of Guided Imagery followed at visit 9. Listen to CDs twice a day 3 days prior to and 2 days following surgery (affect only post surgery outcomes)
  Other Names: Guided Imagery
  Arms: Rest / Guided Imagery

SUMMARY:
The purpose of this study is to determine whether Reiki energy healing affects anxiety and disease progression in patients with localized prostate cancer who are candidates for radical prostatectomy.

DETAILED DESCRIPTION:
120 newly diagnosed prostate cancer patients will be randomized to one of 3 groups: Reiki, another touch therapy, or guided imagery. Subjects in the Reiki and touch therapy groups have 8 sessions in the 4 weeks prior to their medical intervention. Those in the imagery group have one session prior to their medical intervention.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed with prostate cancer
* Scheduled for radial prostatectomy, external beam radiation, brachytherapy, or a combination of these

Exclusion criteria:

* Already involved in energy healing treatments
* Any patient whose medical intervention could not wait the 4-weeks for intervention for medical reasons
* Any patient who gets neo-adjuvant therapy or any herbal product that could affect PSA

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of Reiki on anxiety states using validated psychometric instruments. | Each 30 minute session
To evaluate the effects of Reiki on physiologic anxiety as measured by cortisol and DHEA levels | Each 30 minute session
To evaluate the effects of Reiki on cancer progression as measured by PSA levels in plasma. | throughout study

SECONDARY OUTCOMES:
To evaluate the effects of Reiki and guided imagery on post-surgical pain and urinary symptoms | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Joan Fox, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States